CLINICAL TRIAL: NCT04676451
Title: Femtosecond Laser Assisted Keratotomies for the Management of Corneal Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Seth M Pantanelli, Associate Professor of Ophthalmology, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8058
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Astigmatism; Cataract
Keywords: Astigmatism; Cataract; Femtosecond laser
MeSH Terms: conditions — Astigmatism; Cataract

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, single-arm, interventional clinical trial. Subjects that meet inclusion and exclusion criteria are invited to participate.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Femto-AK Patients (Experimental): Femtosecond laser assisted cataract surgery with creation of astigmatic keratotomies for the correction of corneal astigmatism.
  Interventions: Device: Femto-AK

INTERVENTIONS:
Device: Femto-AK — Astigmatic Keratotomy / Arcuate Incisions for the correction of astigmatism

SUMMARY:
A cataract is a clouding of the lens that occurs naturally with age. Cataract surgery involves removal of the cloudy lens and replacement with an artificial one. A special laser (femtosecond laser) is now being used to help make cataract surgery safer and more accurate . The femtosecond laser can also be used to correct astigmatism, an irregular curvature of the cornea, at the time of cataract surgery through a procedure called astigmatic keratotomy (AK). This study is gathering information about the specific laser settings that are used to perform astigmatic keratotomies (AK) during cataract surgery. This information will be used to improve the outcomes of patients that receive cataract surgery with astigmatic keratotomies in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years of age
* Sex: male or female
* Patients who are planned to undergo femtosecond laser-assisted cataract surgery with astigmatic keratotomy at the Schein Ernst Mishra Eye clinic within the next 60 days of their cataract consultation visit. Subjects with planned single or bilateral cataract eye surgeries are eligible. Planned opposite eye surgery must be within 2-4 weeks of first cataract surgery.
* Fluent in written and spoken English

Exclusion Criteria:

* Patients with corneal dystrophies, including anterior basement membrane dystrophy, keratoconus, and Fuch's endothelial corneal dystrophy.
* Age < 18 years
* Pregnant women
* Cognitive impairment
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Hershey Eye Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- Eyes: Eyes that completed the study
Period: Overall Study
Arm/Group | Eyes
Started | 94; 188 eyes
Completed | 69; 95 eyes
Not Completed | 25; 93 eyes

BASELINE CHARACTERISTICS:
Groups:
- All Participants Who Completed the Study: Ages of all participants
Arm/Group | All Participants Who Completed the Study
Number analyzed (Participants) | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 57
Age, Continuous [Median (Full Range); unit: years] | 73.3734 [57 to 84]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex were not collected from any participant.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Keratometric Correction Index
Description: Keratometric Correction index is the ratio of surgically induced astigmatism to target induced astigmatism. A correction index of 1 suggests that the actual surgically induced astigmatism, as measured by pre- vs- post-op reflectance keratometry, perfectly matched the target (anticipated) induced astigmatism. Correction indices below 1 suggest an under-correction while values above 1 suggest an over-correction.
Time Frame: 1 month
Population: patients underwent cataract extraction with AKs and insertion of a non-toric intraocular lens.
Measure: Mean (Full Range); unit: index
Units Other Than Participants: eyes
Groups:
- Astigmatic Eyes: Eyes with greater than 0.5 D of against-the-rule (ATR) or 1.0 D of with-the-rule (WTR) or oblique (OBL) astigmatism were treated in accordance with the nomogram.
Arm/Group | Astigmatic Eyes
Number analyzed (Participants) | 69
Number analyzed (eyes) | 95
index | 0.51 [0.04 to 3.45]

2. Primary Outcome: Refractive Correction Index
Description: Refractive Correction index is the ratio of surgically induced astigmatism to net effective astigmatism. A correction index of 1 suggests that the actual surgically induced astigmatism, as measured by pre- vs- post-op manifest refraction, perfectly matched the effective astigmatism as estimated by the nomogram. Correction indices below 1 suggest an under-correction while values above 1 suggest an over-correction.
Time Frame: 1 month
Measure: Mean (Full Range); unit: index
Units Other Than Participants: eyes
Arm/Group | Astigmatic Eyes
Number analyzed (Participants) | 69
Number analyzed (eyes) | 95
index | 0.91 [0 to 5.32]

ADVERSE EVENTS:
Time Frame: Adverse events were not captured during the study
Arm/Group | Femto-AK Patients
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT04676451/Prot_SAP_000.pdf